CLINICAL TRIAL: NCT01009034
Title: Study to Determine the Concentrations of Maraviroc in Semen, the Seminal to Plasma Ratio of Maraviroc and the Variability in Seminal to Plasma Ratios Over the Maraviroc Dosing Period.
Brief Title: Concentrations of Maraviroc in the Semen of HIV-Infected Men
Acronym: NCT01009034
Status: Completed | Type: Observational
Sponsor: Canadian Immunodeficiency Research Collaborative (Other)
Responsible Party: Sponsor
Other Study IDs: WS 353380
Record Dates: First submitted 2009-11-05; First posted 2009-11-06 (Estimated); Results first posted 2014-09-09 (Estimated); Last update posted 2014-09-09 (Estimated); Status verified 2014-09

CONDITIONS: Maraviroc Concentrations in Semen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 12 male HIV-positive patients: Male HIV-positive patients who have been receiving stable antiretroviral therapy that includes maraviroc for a minimum of three months.
  Interventions: Other: Measuring semen samples

INTERVENTIONS:
Other: Measuring semen samples — Measure semen sample concentrations, obtain semen to plasma ratios across the dosing interval, the area under the concentration time curve of maraviroc in semen, the variability in the penetration of maraviroc into the seminal compartment over the raltegravir dosing period.

SUMMARY:
The objective of this study is to determine if concentrations of maraviroc in semen exceed the 50% and 95% inhibitory concentrations of HIV during the dose interval.

The secondary objective is to determine the extent of maraviroc penetration into semen by obtaining semen to plasma ratios across the dosing interval, to determine the area under the concentration time curve of maraviroc in semen, and to determine the variability in the penetration of maraviroc into the seminal compartment over the maraviroc dosing period.

DETAILED DESCRIPTION:
The patient population will consist of 12 male HIV-positive patients who have been receiving stable antiretroviral therapy that includes maraviroc for a minimum of three months. Patients will be enrolled from one clinic in downtown Toronto and a hospital affiliated HIV specialty clinic in Ottawa, Ontario. Eligible patients will have evidence of full virologic suppression (HIV viral load < 50 copies/mL) at least one month prior to enrollment in the study. No changes will be made to the patients antiretroviral therapy during the course of the study.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected male
* 18 years old or older
* on maraviroc twice daily as part of their antiretroviral regimen for at least 3 months prior to screening
* viral load < 50 copies/mL at least one month prior to enrolling
* able to read, understand and sign a written informed consent prior to initiation of the study
* medically stable at the time of the study, with no evidence of acute illness

Exclusion Criteria:

* having difficulty adhering to current antiretroviral therapy
* patient is expected to have difficulties adhering with study protocol
* patients with malignancy, or acute renal or liver disease
* patient with active AIDS-defining illness
* patient with any medical, psychiatric or other circumstance that may impede the provision of informed consent
* patient with any of the following abnormalities at the time of screening:
* hemoglobin < 85 g/L
* absolute neutrophil count < 1000 cells/uL
* platelet count < 50,000 cells/uL
* AST, ALT or total bilirubin > 3 times the upper limit of normal
* serum creatinine > 1.5 times upper limit of normal
* patient receiving concomitant therapy with rifampin or St. John's wort

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 12 HIV-positive males
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2009-10; Primary Completion 2011-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - The Ottawa Hospital, Ottawa, Ontario
  - Canadian Immunodeficiency Research Collaborative, Toronto, Ontario

RESULTS

PARTICIPANT FLOW:
Groups:
- 10 Male HIV-positive Patients: Male HIV-positive patients who have been receiving stable antiretroviral therapy that includes maraviroc for a minimum of three months.
  Measuring semen samples: Measure semen sample concentrations, obtain semen to plasma ratios across the dosing interval, the area under the concentration time curve of maraviroc in semen, the variability in the penetration of maraviroc into the seminal compartment over the raltegravir dosing period.
Period: Overall Study
Arm/Group | 10 Male HIV-positive Patients
Started | 14
Completed | 10
Not Completed | 4
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: 10 HIV+ men on maraviroc with VL <50 copies per M
Arm/Group | 10 Male HIV-positive Patients
Number analyzed (Participants) | 14
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 51 [46 to 57]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 14
Region of Enrollment [Number; unit: participants]
  Canada | 14

OUTCOME MEASURES:

1. Primary Outcome: Semen to Plasma Ratio of HIV Concentration During the Dosing Interval for Dar, Evr, Mar & Ral.
Description: We used a staggered sampling approach in which semen samples were produced by participants over several days at different sampling times relative to the morning dose of antiretrovirals. Speciﬁ- cally, semen samples were collected 30 minutes to 1 hour before the morning dose of medication (day 1), and then at hours 1, 2, 4, 8, and 12 postdrug ingestion on days 2-6. We collected corresponding blood samples within 1 hour of the semen sample. For each participant a single value (the HIV concentration ratio) was calculated as the minimum HIV concentration in the semen over the minimum HIV concentration in the blood throughout the dosing interval.
Time Frame: Semen samples were collected 30 minutes to 1 hour before the morning dose of medication (day 1), and then at hours 1, 2, 4, 8, and 12 postdrug ingestion on days 2-6. Blood samples were collected within 1 hour of the semen sample.
Population: We used a staggered sampling approach in which semen samples were produced by participants over several days at different sampling times relative to the morning dose of antiretrovirals.
Measure: Median (Inter-Quartile Range); unit: Inhibitory concentration ratio
Arm/Group | 10 Male HIV-positive Patients
Number analyzed (Participants) | 10
Inhibitory concentration ratio
  dar | 0.20 [0.14 to 0.24]
  evr | 0.16 [0.15 to 0.23]
  mar | 0.92 [0.59 to 1.91]
  ral | 4.32 [4.1 to 5.0]

2. Secondary Outcome: Determine the Extent of Maraviroc Penetration Into Semen by Obtaining Semen to Plasma Ratios Across the Dosing Interval
Description: For each participant, the Maraviroc penetration ratio was calculated as the maximum Maraviroc concentration in the semen over the maximum Maraviroc concentration in the blood throughout the dosing interval.
Time Frame: as for outcome 1
Measure: Mean (Inter-Quartile Range); unit: ratio
Arm/Group | 10 Male HIV-positive Patients
Number analyzed (Participants) | 10
ratio | 0.62 [0.23 to 2.45]

3. Secondary Outcome: Determine the Area Under the Concentration Time Curve of Maraviroc in Semen.
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: h*mg/L
Arm/Group | 10 Male HIV-positive Patients
Number analyzed (Participants) | 10
h*mg/L | 3.43 [1.83 to 7.96]

ADVERSE EVENTS:
Arm/Group | 12 Male HIV-positive Patients
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days